CLINICAL TRIAL: NCT02187055
Title: A Phase 3b/4 Randomized Double Blind Study Of 5 Mg Of Tofacitinib With And Without Methotrexate In Comparison To Adalimumab With Methotrexate In Subjects With Moderately To Severely Active Rheumatoid Arthritis
Brief Title: An Efficacy And Safety Study Evaluating Tofacitinib With And Without Methotrexate Compared To Adalimumab With Methotrexate
Acronym: ORAL STRATEGY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921187; 2014-000358-13 (EudraCT Number); ORAL STRATEGY (Other: Alias Study Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Rhematoid Arthritis
MeSH Terms: interventions — tofacitinib; Methotrexate; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tofacitinib 5 mg twice daily with methotrexate (Experimental)
  Interventions: Drug: Tofacitinib with methotrexate
- Tofacitinib 5 mg twice daily monotherapy (Experimental)
  Interventions: Drug: Tofacitinib without methotrexate
- Adalimumab with methotrexate (Active Comparator)
  Interventions: Biological: Adalimumab with methotrexate

INTERVENTIONS:
Drug: Tofacitinib with methotrexate — Tofacitinib 5 mg twice daily, oral for 12 months Methotrexate (previous stable dose 15-25 mg) every week, oral for 12 months Placebo for adalimumab every other week, subcutaneous for 12 months
  Arms: Tofacitinib 5 mg twice daily with methotrexate
Drug: Tofacitinib without methotrexate — Tofacitinib 5 mg twice daily, oral for 12 months Placebo for methotrexate (previous stable dose) every week, oral for 12 months Placebo for adalimumab every other week, subcutaneous for 12 months
  Arms: Tofacitinib 5 mg twice daily monotherapy
Biological: Adalimumab with methotrexate — Placebo for tofacitinib twice daily, oral for 12 months Methotrexate (previous stable dose 15-25 mg) every week, oral for 12 months Adalimumab 40 mg every other week, subcutaneous for 12 months
  Arms: Adalimumab with methotrexate

SUMMARY:
To assess the efficacy of tofacitinib monotherapy or tofacitinib with methotrexate as compared to adalimumab with methotrexate. To compare the efficacy of tofacitinib monotherapy compared to tofacitinib combined with methotrexate. To compare effects on all health outcomes measures in the study. To evaluate the safety and tolerability of tofacitinib and adalimumab. To evaluate the safety of the zoster vaccine given prior to the initiation of tofacitinb or adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe rheumatoid arthritis
* On methotrexate but inadequately controlled
* Subjects must not have active tuberculosis or an inadequately treated tuberculosis infection
* Subjects must use contraception

Exclusion Criteria:

* Subjects who have been previously treated with adalimumab or Tofacitinib
* Subjects with any current malignancy or a history of malignancy, with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Subjects with specific laboratory test abnormalities
* Subjects with specific types of infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (215):
- United States (60):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arthrocare, Arthritis Care & Research, PC, Gilbert, Arizona
  - Medvin Clinical Research, Covina, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - HealthCare Partners Medical Group, Huntington Beach, California
  - Keck Medicine of USC - Division of Rheumatology, Los Angeles, California
  - University of Southern California (USC) Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center - Drug Information Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California
  - Medvin Clinical Research, Placentia, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Medvin Clinical Research, Van Nuys, California
  - Medvin Clinical Research, Whittier, California
  - Joao M. A. Nascimento, Bridgeport, Connecticut
  - AARDS Research, Inc., Aventura, Florida
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Gulf Region Clinical Research Institute Llc, Pensacola, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - BayCare Medical Group Inc, Tampa, Florida
  - The Center for Arthritis and Rheumatism, Vero Beach, Florida
  - The Office of Alastair C. Kennedy, MD, Vero Beach, Florida
  - Advanced Clinical Research of Orlando, Inc., Winter Garden, Florida
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Diagnostic Rheumatology and Research PC, Indianapolis, Indiana
  - Ochsner Clinic Baton Rouge, Baton Rouge, Louisiana
  - Arthritis and Diabetes Clinic, Inc, Monroe, Louisiana
  - Arthritis Treatment Center, Frederick, Maryland
  - Jasper Clinic, Kalamazoo, Michigan
  - Arthritis and Osteoporosis Treatment and Research Center, Flowood, Mississippi
  - Clinvest/ A Division of Banyan Group, Inc., Springfield, Missouri
  - St. Louis Center For Clinical Research Barbara Caciolo, MD, St Louis, Missouri
  - Dr. Prem C. Chatpar M.D.,LLC, Plainview, New York
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Rowan Diagnostic Clinic, Salisbury, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Trinity Health Center - Medical Arts, Minot, North Dakota
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Arthritis Care And Diagnostic Center, P.A., Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
  - Rheumatology Clinic of Houston, PA, Houston, Texas
  - Houston Institute For Clinical Research, Houston, Texas
  - Arthritis & Osteoporosis Associates, LLP, Lubbock, Texas
  - Southwest Rheumatology Research, LLC., Mesquite, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (5):
  - Atencion Integral en Reumatologia (AIR), CABA, Buenos Aires
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro Radiologico Luis Mendez Collado SRL, San Miguel de Tucumán, Tucumán Province
  - Organizacion Medica de Investigacion S.A - OMI, Buenos Aires
  - CER San Juan, Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Pacific Private Clinic, Southport, Queensland
  - QML Pathology, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Emeritus Research, Malvern East, Victoria
  - RK Will Pty Ltd, Victoria Park, Western Australia
- Bosnia and Herzegovina (2):
  - University Hospital Clinical Center Banja Luka, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla, Tuzla
- Bulgaria (9):
  - UMHAT "Dr. Georgi Stranski" EAD, Pleven
  - MHAT "Kaspela" EOOD, Plovdiv
  - MHAT EUROHOSPITAL Plovdiv, Plovdiv
  - MHAT Akta Medika OOD, Rousse
  - MHAT Ruse AD, Rousse
  - MHAT Shumen AD, Shumen
  - NMTH Tsar Boris Clinic of Internal Diseases, Sofia
  - MHAT Lyulin EAD, Sofia
  - MHAT "Targovishte" AD, Targovisthe
- Canada (2):
  - Kw Musculoskeletal Research Inc, Kitchener, Ontario
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Chile (4):
  - Quantum Research Ltda, Puerto Varas, Los Lagos Region
  - Quantum Research, Puerto Varas, Los Lagos Region
  - Estudios Clinicos Quinta Region Ltda., Viña del Mar, Región de Valparaíso
  - Prosalud, Santiago, Santiago Metropolitan
- Czechia (5):
  - Revmacentrum MUDr. Mostera, s.r.o., Brno-Židenice, Czech Republic
  - Revmatologie s.r.o., Brno
  - Revmatologicka ambulance, Česká Lípa
  - Vesalion, s.r.o., Ostrava- Moravska Ostrava
  - Revmatologie, Prague
- Estonia (3):
  - Foundation Parnu Hospital, Pärnu
  - East-Tallinn Central Hospital Ltd, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Latvia (2):
  - Health Center 4, Riga
  - ORTO clinic Ltd, Riga
- Lithuania (3):
  - Alytaus District S. Kudirkos Hospital, Alytus
  - VAKK "Clinic of Dr. Kilda", Kaunas
  - PI Republican Siauliai Hospital, Šiauliai
- Mexico (13):
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas S. C., Torreón, Coahuila
  - Centro Integral en Reumatologia, SA de CV, Guadalajara, Jalisco
  - CINTRE, Centro de Investigacion y Tratamiento Reumatologico S.C. Consultorio Medico de Reumatologia, Mexico City, Mexico City
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa S.C., Culiacán, Sinaloa
  - Centro de Investigacion en Tratamientos Innovadores de Sinaloa S.C., Culiacán, Sinaloa
  - Centro Multidisciplinario para el Desarrollo Especializado de la Invetigacion Clinica en Yucatan, Mérida, Yucatán
  - Departamento de Imagen de Hospital Star Medica Merida, Mérida, Yucatán
  - Laboratorio clínico del Hospital Star Medica Merida, Mérida, Yucatán
  - Storage for lab kits and study materials, Mérida, Yucatán
  - Investigacion y Biomedica de Chihuahua, SC, Chihuahua City
  - Centro de Integral en Reumatologia SA de CV, Jalisco
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, S.C., San Luis Potosí City
  - Unidad de Investigaciones Reumatologicas A.C., San Luis Potosí City
- Peru (4):
  - Unidad de Investigacion en Medicina Interna y Enfermedades criticas-Hogar Clinica San Juan de Dios, Arequipa
  - ABK REUMAR S.R.L. de Medicentro Biociencias_ BIO CIENCIAS PERU S.R.L., Lima
  - Instituto Peruano del Hueso y la Articulacion, Lima
  - Investigaciones Clinicas S.A.C., Lima
- Philippines (10):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Brokenshire Integrated Health Ministries, Inc., Davao City, Davao DEL SUR
  - Iloilo Doctors' Hospital, Inc, Iloilo City, Iloilo
  - University of the Philippines Manila-Philippine General Hospital, Manila, National Capital Region
  - Jose R. Reyes Memorial Medical Center-Rayuma Klinik, Manila, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Far Eastern University - NRMF Medical Center, Quezon City, National Capital Region
  - Perpetual Succour Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City
- Poland (14):
  - Medica Pro Familia Sp. z o.o. S.K.A. Oddzial Krakow, Krakow, Malopolska
  - Centrum Medyczne Amed, Warsaw, WOJ Mazowieckie
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy,, Bydgoszcz
  - Centrum Medyczne SILESIANA Sp. z o.o., Bytom
  - Nzoz Bif-Med, Bytom
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka, Elblag
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Lecznica MAK-MED, NZOZ, Nadarzyn
  - Prywatna Praktyka Lekarska, Poznan
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
- Romania (11):
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca Reumatologie, Cluj-Napoca, Cluj
  - Covamed Serv SRL, Sfântu Gheorghe, Covasna
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris", Baia Mare, Maramureş
  - S.C. Clinica Somesan S.R.L., Baia Mare, Maramureş
  - Ianuli Med Consult SRL, Reumatologie, Bucharest
  - Spitalul Clinic Sf. Maria, Medicina interna - Reumatologie, Bucharest
  - Spitalul Clinic Sf. Maria, Bucharest
  - Spitalul Clinic "Dr. I. Cantacuzino", Bucharest
  - Centrul Clinic de Boli Reumatismale "Dr. Ion Stoia", Bucharest
  - Spitalul Clinic Judetean de Urgenta - "Sf.Apostol Andrei" Galati, Galati
  - Spitalul Clinic de Recuperare Iasi, Iași
- Russia (14):
  - Republic Hospital n.a. V.A. Baranov, Petrozavodsk, Karelia Republic
  - State Budgetary Healthcare Institution of Karelia Republic "Republic Hospital n.a. V.A. Baranov", Petrozavodsk, Karelia Republic
  - SAHI of KR "Kemerovo Regional Clinical Hospital", Kemerovo
  - SBEI HPE First Moscow State Medical University n.a.I.M.Sechenov of MoH of RF based on UCH#1, Moscow
  - CJSC "European Medical Center", Moscow
  - SBEI HPE Novosibirsk State Medical University of MoH of RF, Novosibirsk
  - State Budgetary Healthcare Institution "Orenburg Regional Clinical Hospital", Orenburg
  - State Budgetary Institution of Ryazan Region "Regional Clinical Cardiology Dispensary", Ryazan
  - Limited Liability Company AVA-PETER, Saint Petersburg
  - State Budgetary Institution of Healthcare "Samara Regional Clinical Hospital n.a. V.D. Seredavin", Samara
  - State Institution of Healthcare "Regional Clinical Hospital", Saratov
  - Non-state Healthcare Institution "Regional Hospital at Smolensk Station of OJSC "Russian Railways", Smolensk
  - State Autonomous Healthcare lnstitution of Yarostavl Region, Yaroslavl
  - State Budgetary Healthcare Institution of Yaroslavl Region "Clinical Hospital #3", Yaroslavl
- South Africa (12):
  - Iatros International, Bloemfontein, Free State
  - LCS Clinical Research Unit, Johannesburg, Gauteng
  - WCR: Wits Clinical Research Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - WCR: Wits Clinical Research, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
  - Clinical Research Unit, University of Pretoria, Pretoria, Gauteng
  - Netcare Jakaranda Hospital, Pretoria, Gauteng
  - University of Pretoria, Pretoria, Gauteng
  - Netcare St Augustine's Hospital, Durban, KwaZulu-Natal
  - Arthritis Clinical Research Trials, Cape Town, Western Cape
  - Panorama Medical Centre, Cape Town, Western Cape
  - Wineland Medical Research Centre, Stellenbosch, Western Cape
- South Korea (6):
  - Inha University Hospital, Jung-Gu, Incheon
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Infanta Luisa, Seville
- Taiwan (6):
  - Chung Shan Medical University Hospital, Taichung, Taiwan ROC
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital - New, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan
- Thailand (5):
  - Phramongkutklao Hospital, Bangkok, Rajthevi
  - Cardiology Unit,Department of Medicine, Faculty of Medicine, Ramathibodi Hospital,Mahidol University, Bangkok
  - Div. of Allergy Immunology and Rheumatology, Dept. of Medicine,, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Songklanagarind Hospital - Prince of Songkhla University, Songkhla
- Turkey (Türkiye) (4):
  - Ankara Universitesi Tip Fakultesi Ibn-i Sina Hastanesi, Ankara
  - Ondokuz Mayis Universitesi Tip Fakultesi Saglik Uyg. ve Eg., Samsun
  - Ondokuz Mayis Universitesi Tip Fakultesi Saglik Uygulama ve Egitim Merkezi, Samsun
  - Cumhuriyet Universitesi Tip Fakultesi Hastanesi, Sivas
- United Kingdom (5):
  - The Dudley Group NHS Foundation Trust, Dudley, WEST Midlands
  - The Royal Wolverhamptons NHS Trust, Cannock
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal Free London NHS Foundation Trust, London

REFERENCES:
- [Derived] Takeuchi T, Tanaka Y, Yamanaka H, Yamaoka K, Sugiyama N, Iikuni N, Toyoizumi S, Kwok K, Tsai WC, Mysler E, Moots RJ, Smolen JS, Fleischmann R. Efficacy and Safety of Tofacitinib and Adalimumab in Rheumatoid Arthritis by Body Mass Index-Normalized Methotrexate Dose: A Post Hoc Analysis. Rheumatol Ther. 2026 Jan 22. doi: 10.1007/s40744-025-00823-0. Online ahead of print. PMID 41565911
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Pope J, Finckh A, Silva-Fernandez L, Mandl P, Fan H, Rivas JL, Valderrama M, Montoro M. Tofacitinib Monotherapy in Rheumatoid Arthritis: Clinical Trials and Real-World Data Contextualization of Patients, Efficacy, and Treatment Retention. Open Access Rheumatol. 2024 Jun 11;16:115-126. doi: 10.2147/OARRR.S446431. eCollection 2024. PMID 38883150
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Bessette L, Mysler E, Kinch CD, Kwok K, Lukic T, On PV, van Vollenhoven RF. Impact of Tofacitinib on Components of the ACR Response Criteria: Post Hoc Analysis of Phase III and Phase IIIb/IV Trials. J Rheumatol. 2022 Jun;49(6):566-576. doi: 10.3899/jrheum.210707. Epub 2022 Mar 1. PMID 35232809
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Takeuchi T, Fleischmann R, Iikuni N, Shi H, Soma K, Paulissen J, Hirose T, Smolen JS. Differences and similarities in clinical and functional responses among patients receiving tofacitinib monotherapy, tofacitinib plus methotrexate, and adalimumab plus methotrexate: a post hoc analysis of data from ORAL Strategy. Arthritis Res Ther. 2021 Aug 24;23(1):220. doi: 10.1186/s13075-021-02591-y. PMID 34429160
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Strand V, Mysler E, Moots RJ, Wallenstein GV, DeMasi R, Gruben D, Soma K, Iikuni N, Smolen JS, Fleischmann R. Patient-reported outcomes for tofacitinib with and without methotrexate, or adalimumab with methotrexate, in rheumatoid arthritis: a phase IIIB/IV trial. RMD Open. 2019 Oct 1;5(2):e001040. doi: 10.1136/rmdopen-2019-001040. eCollection 2019. PMID 31673419
- [Derived] Calabrese LH, Abud-Mendoza C, Lindsey SM, Lee SH, Tatulych S, Takiya L, Iikuni N, Soma K, Luo Z, Fleischmann R. Live Zoster Vaccine in Patients With Rheumatoid Arthritis Treated With Tofacitinib With or Without Methotrexate, or Adalimumab With Methotrexate: A Post Hoc Analysis of Data From a Phase IIIb/IV Randomized Study. Arthritis Care Res (Hoboken). 2020 Mar;72(3):353-359. doi: 10.1002/acr.24010. PMID 31207152
- [Derived] Fleischmann R, Mysler E, Hall S, Kivitz AJ, Moots RJ, Luo Z, DeMasi R, Soma K, Zhang R, Takiya L, Tatulych S, Mojcik C, Krishnaswami S, Menon S, Smolen JS; ORAL Strategy investigators. Efficacy and safety of tofacitinib monotherapy, tofacitinib with methotrexate, and adalimumab with methotrexate in patients with rheumatoid arthritis (ORAL Strategy): a phase 3b/4, double-blind, head-to-head, randomised controlled trial. Lancet. 2017 Jul 29;390(10093):457-468. doi: 10.1016/S0140-6736(17)31618-5. Epub 2017 Jun 16. PMID 28629665
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921187&StudyName=An%20Efficacy%20And%20Safety%20Study%20Evaluating%20Tofacitinib%20With%20And%20Without%20Methotrexate%20Compared%20To%20Adalimumab%20With%20Methotrexate

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although a total of 1,152 participants were randomized, only 1,146 participants received treatment and are included in the full analysis set summarized below.
Groups:
- Tofacitinib 5 mg BID: One active tofacitinib 5 mg tablet orally BID plus placebo MTX (prior dose) orally every week plus placebo adalimumab 40 mg subcutaneously (SC) every other week for up to 12 months.
- Tofacitinib 5 mg BID + MTX: One active tofacitinib 5 mg tablet orally BID plus active MTX (prior dose) orally every week plus placebo adalimumab 40 mg SC every other week for up to 12 months.
- Adalimumab 40 mg + MTX: One placebo tofacitinib 5 mg tablet orally BID plus active MTX (prior dose) orally every week plus active adalimumab 40 mg SC every other week for up to 12 months.
Period: Overall Study
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Started | 384 (Treated) | 376 (Treated) | 386 (Treated)
Completed | 315 | 303 | 312
Not Completed | 69 | 73 | 74
Not completed — Lack of Efficacy | 10 | 3 | 7
Not completed — Lost to Follow-up | 2 | 7 | 3
Not completed — No longer meets eligibility criteria | 0 | 2 | 0
Not completed — No longer willing to participate | 6 | 8 | 10
Not completed — Other | 5 | 6 | 3
Not completed — Protocol Violation | 9 | 9 | 4
Not completed — Pregnancy | 3 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 11 | 11
Not completed — Adverse Event | 21 | 26 | 36
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX | Total
Number analyzed (Participants) | 384 | 376 | 386 | 1146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (12.2) | 50.0 (13.4) | 50.7 (13.4) | 50.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 311 | 320 | 950
  Male | 65 | 65 | 66 | 196

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology Criteria 50% Improvement (ACR50) Response at Month 6
Description: ACR50 is a greater than or equal to (≥) 50 percent (%) improvement in tender joint count (TJC) or swollen joint count (SJC) and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment (PGA) of disease activity, 2) participant's assessment (PtGA) of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein (CRP) at each visit.
Time Frame: Month 6
Population: Full analysis set (FAS) included all participants who were randomized and received at least one dose of the randomized investigational drug (tofacitinib or adalimumab).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 384 | 376 | 386
Percentage of participants | 38.28 | 46.01 | 43.78
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Non-Inferiority or Equivalence — Non-inferiority was a treatment difference larger than -13% at the population level; p = 0.2101, Normal approximation to proportions; Multiplicity-adjusted; Difference in response rate = -7.73, 98.34% CI 2-sided [-16.29 to 0.83]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Non-Inferiority or Equivalence — Non-inferiority was a treatment difference larger than -13% at the population level; p = 0.0512, Normal approximation to proportions; Multiplicity-adjusted; Difference in response rate = -5.50, 98.34% CI 2-sided [-13.98 to 2.98]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Non-Inferiority or Equivalence — Non-inferiority was a treatment difference larger than -13% at the population level; p < 0.0001, Normal approximation to proportions; Multiplicity adjusted; Difference in response rate = 2.23, 98.34% CI 2-sided [-6.40 to 10.86]

2. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Value at Month 6
Description: SDAI is the numerical sum of five outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 centimeter (cm) visual analogue scale (VAS) (higher scores indicate greater affection due to disease activity), and CRP (mg/dL). SDAI total score ranges from 0 to 86. SDAI less than or equal to (≤) 3.3 indicates disease remission, >3.4 to 11 indicates low disease activity, >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 355 | 343 | 345
Score on a scale | -23.7 (0.62) | -26.6 (0.62) | -25.6 (0.62)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = 2.8, 95% CI 2-sided [1.23 to 4.41]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.9, 95% CI 2-sided [0.33 to 3.49]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.9, 95% CI 2-sided [-2.51 to 0.68]

3. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Value at Month 6
Description: CDAI is the numerical sum of four outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity). CDAI total score ranges from 0 to 76. CDAI ≤2.8 indicates disease remission, >2.8 to 10 indicates low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicates high disease activity.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 345 | 347
Score on a scale | -22.9 (0.61) | -25.5 (0.61) | -24.8 (0.61)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = 2.6, 95% CI 2-sided [1.08 to 4.18]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.9, 95% CI 2-sided [0.40 to 3.48]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.7, 95% CI 2-sided [-2.24 to 0.86]

4. Secondary Outcome: Change From Baseline in Disease Activity Score 28-4 (DAS28-4) Including CRP at Month 6
Description: DAS28-4 (CRP) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and CRP (mg/L) using the following: DAS28-4(CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014* PtGA (millimeters [mm]) + 0.96. Total score range: 0 to 9.4, higher score indicated higher disease activity. DAS28-4 (CRP) ≤3.2 indicates low disease activity, >3.2 to 5.1 indicates moderate to high disease activity, and less than (<) 2.6 indicates remission.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 355 | 343 | 345
Score on a scale | -2.1 (0.07) | -2.5 (0.07) | -2.3 (0.07)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [0.16 to 0.50]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.2, 95% CI 2-sided [0.05 to 0.39]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.1, 95% CI 2-sided [-0.28 to 0.06]

5. Secondary Outcome: Change From Baseline in Disease Activity Score 28-4 (DAS28-4) Including Erythrocyte Sedimentation Rate (ESR) at Month 6
Description: DAS28-4 (ESR) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and ESR (mm/hour) using the following: DAS28-4(ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014* PtGA (mm). Total score range: 0 to 9.4, higher score indicated higher disease activity. DAS28-3 (ESR) ≤3.2 indicates low disease activity, >3.2 to 5.1 indicates moderate to high disease activity, and <2.6 indicates remission.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 349 | 342 | 343
Score on a scale | -2.1 (0.07) | -2.4 (0.07) | -2.4 (0.07)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [0.15 to 0.51]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [0.10 to 0.46]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.0, 95% CI 2-sided [-0.23 to 0.13]

6. Secondary Outcome: Percentage of Participants Achieving Observed American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) Boolean Remission Criteria at Month 6
Description: To meet the ACR-EULAR Boolean remission criteria, a participant must satisfy all of the following: TJC ≤1 and SJC ≤1 (both based on a 28-joint assessment), CRP ≤1 mg/dL, and PtGA ≤1 on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity).
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 358 | 346 | 355
Percentage of participants | 7.54 | 8.67 | 9.58
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in remission rate = -1.21, 95% CI 2-sided [-4.99 to 2.56]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -1.78, 95% CI 2-sided [-5.59 to 2.04]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -0.56, 95% CI 2-sided [-4.53 to 3.40]

7. Secondary Outcome: Percentage of Participants Achieving SDAI ≤3.3 at Month 6
Description: SDAI is the numerical sum of five outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity), and CRP (mg/dL). SDAI total score ranges from 0 to 86. SDAI ≤3.3 indicates disease remission.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 345 | 348
Percentage of participants | 10.64 (0.62) | 13.91 (0.62) | 14.37 (0.62)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in remission rate = -3.40, 95% CI 2-sided [-7.95 to 1.15]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -3.06, 95% CI 2-sided [-7.55 to 1.43]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = 0.34, 95% CI 2-sided [-4.45 to 5.14]

8. Secondary Outcome: Percentage of Participants Achieving CDAI ≤2.8 at Month 6
Description: CDAI is the numerical sum of four outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity). CDAI total score ranges from 0 to 76. CDAI ≤2.8 indicates disease remission.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 358 | 347 | 350
Percentage of participants | 10.89 | 14.70 | 14.57
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in remission rate = -3.67, 95% CI 2-sided [-8.29 to 0.94]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -3.06, 95% CI 2-sided [-7.59 to 1.48]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = 0.62, 95% CI 2-sided [-4.24 to 5.47]

9. Secondary Outcome: Percentage of Participants Achieving DAS28-4 (ESR) <2.6 at Month 6
Description: DAS28-4 (ESR) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and ESR (mm/hour) using the following: DAS28-4(ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014* PtGA (mm). Total score range: 0 to 9.4, higher score indicates higher disease activity. DAS28-4 (ESR) <2.6 indicates disease remission.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 353 | 344 | 346
Percentage of participants | 11.33 | 12.79 | 13.58
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in remission rate = -1.55, 95% CI 2-sided [-6.03 to 2.93]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -2.02, 95% CI 2-sided [-6.51 to 2.47]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -0.47, 95% CI 2-sided [-5.11 to 4.18]

10. Secondary Outcome: Percentage of Participants Achieving DAS28-4 (CRP) <2.6 at Month 6
Description: DAS28-4 (CRP) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and CRP (mg/L) using the following: DAS28-4(CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014* PtGA (mm) + 0.96. Total score range: 0 to 9.4, higher score indicates higher disease activity. DAS28-4 (CRP) <2.6 indicates remission.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 345 | 348
Percentage of participants | 22.69 | 32.75 | 30.17
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in remission rate = -9.49, 95% CI 2-sided [-15.68 to -3.30]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = -6.89, 95% CI 2-sided [-12.94 to -0.83]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in remission rate = 2.61, 95% CI 2-sided [-3.86 to 9.07]

11. Secondary Outcome: Percentage of Participants Achieving SDAI ≤11 at Month 6
Description: SDAI is the numerical sum of five outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity), and CRP (mg/dL). SDAI total score ranges from 0 to 86. SDAI ≤3.3 indicates disease remission, >3.4 to 11 indicates low disease activity.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 345 | 348
Percentage of participants | 46.78 (0.62) | 53.33 (0.62) | 51.15 (0.62)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -6.24, 95% CI 2-sided [-13.32 to 0.84]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -3.66, 95% CI 2-sided [-10.69 to 3.37]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = 2.58, 95% CI 2-sided [-4.51 to 9.68]

12. Secondary Outcome: Percentage of Participants Achieving CDAI ≤10 at Month 6
Description: CDAI is the numerical sum of four outcome parameters: TJC and SJC both based on a 28-joint assessment, PtGA and PGA both assessed on a 0 to 10 cm VAS (higher scores indicate greater affection due to disease activity). CDAI total score ranges from 0 to 76. CDAI ≤2.8 indicates disease remission, >2.8 to 10 indicates low disease activity.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 358 | 347 | 350
Percentage of participants | 45.53 | 52.45 | 50.00
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -6.22, 95% CI 2-sided [-13.29 to 0.85]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -3.93, 95% CI 2-sided [-10.94 to 3.09]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = 2.30, 95% CI 2-sided [-4.79 to 9.39]

13. Secondary Outcome: Percentage of Participants Achieving DAS28-4 (ESR) ≤3.2 at Month 6
Description: DAS28-4 (ESR) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and ESR (mm/hour) using the following: DAS28-4(ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014* PtGA (mm). Total score range: 0 to 9.4, higher score indicates higher disease activity. DAS28-4 (ESR) ≤3.2 indicates low disease activity.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 353 | 344 | 346
Percentage of participants | 22.10 | 28.49 | 29.77
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -6.02, 95% CI 2-sided [-12.05 to 0.00]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -6.89, 95% CI 2-sided [-12.90 to -0.87]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -0.87, 95% CI 2-sided [-7.17 to 5.44]

14. Secondary Outcome: Percentage of Participants Achieving DAS28-4 (CRP) ≤3.2 at Month 6
Description: DAS28-4 (CRP) was calculated from the SJC and TJC (both based on a 28-joint assessment), PtGA (assessed on a 0 to 10 cm VAS; higher scores indicate greater affection due to disease activity) and CRP (mg/L) using the following: DAS28-4(CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014* PtGA + 0.96. Total score range: 0 to 9.4, higher score indicated higher disease activity. DAS28-4 (CRP) ≤3.2 indicates low disease activity.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 345 | 348
Percentage of participants | 44.54 | 49.57 | 50.86
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -4.87, 95% CI 2-sided [-11.92 to 2.18]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -5.48, 95% CI 2-sided [-12.49 to 1.52]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in rresponse rate = -0.61, 95% CI 2-sided [-7.70 to 6.47]

15. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology Criteria 20% Improvement (ACR20) Response at Month 6
Description: ACR20 response is a ≥20% improvement in TJC or SJC and 20% improvement in 3 of the following 5 criteria: 1) PGA of disease activity, 2) PtGA of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 354 | 345 | 349
Percentage of participants | 70.06 | 79.13 | 77.65
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -8.29, 95% CI 2-sided [-14.84 to -1.75]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -6.14, 95% CI 2-sided [-12.72 to 0.44]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = 2.15, 95% CI 2-sided [-4.22 to 8.52]

16. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology Criteria 70% Improvement (ACR70) Response at Month 6
Description: ACR70 response is a ≥70% improvement in TJC or SJC and 70% improvement in 3 of the following 5 criteria: 1) PGA of disease activity, 2) PtGA of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 343 | 349
Percentage of participants | 19.66 | 27.11 | 22.64
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; Difference in response rate = -6.77, 95% CI 2-sided [-12.61 to -0.93]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -2.50, 95% CI 2-sided [-8.09 to 3.10]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = 4.27, 95% CI 2-sided [-1.68 to 10.23]

17. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Month 6
Description: The HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dressing and grooming, arising, eating, walking, reach, grip, hygiene and other activities over the past week. Each activity category consists of 2 to 3 items. Each item is scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity requiring assistance from another individual or the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 348 | 350
Units on a scale | -0.52 (0.031) | -0.58 (0.031) | -0.54 (0.031)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = 0.07, 95% CI 2-sided [-0.011 to 0.148]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.03, 95% CI 2-sided [-0.054 to 0.105]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.04, 95% CI 2-sided [-0.122 to 0.037]

18. Secondary Outcome: Percentage of Participants Achieving an HAQ-DI Decrease of at Least 0.22 at Month 6
Description: The HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dressing and grooming, arising, eating, walking, reach, grip, hygiene and other activities over the past week. Each activity category consists of 2 to 3 items. Each item is scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity requiring assistance from another individual or the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. A decrease of 0.22 or more is considered a positive response.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 348 | 350
Percentage of participants | 71.07 | 75.57 | 72.86
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -4.07, 95% CI 2-sided [-10.68 to 2.55]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = -1.21, 95% CI 2-sided [-7.87 to 5.44]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; Difference in response rate = 2.86, 95% CI 2-sided [-3.72 to 9.43]

19. Secondary Outcome: Change From Baseline in the Short-Form-36 (SF-36) Health Survey, Physical Component Score at Month 6
Description: The SF-36 health survey is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The health domains are aggregated into two summary scores known as the physical component summary (PCS) score and the mental component summary (MCS) score. Normalized domain scores, PCS and MCS scores are used in the analyses. The component and domain scores were scored using the United States (US) 1998 general population norms. The resulting norm-based scores for both the SF-36 version 2 (v2) and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher PCS score represents better physical health status.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 355 | 346 | 349
Score on a scale | 6.7 (0.44) | 7.9 (0.43) | 7.8 (0.43)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -1.2, 95% CI 2-sided [-2.28 to -0.11]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -1.1, 95% CI 2-sided [-2.16 to 0.01]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.1, 95% CI 2-sided [-0.97 to 1.20]

20. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Mental Component Score at Month 6
Description: The SF-36 health survey is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The health domains are aggregated into two summary scores known as the PCS score and the MCS score. Normalized domain scores, PCS and MCS scores are used in the analyses. The component and domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher MCS score represents better physical health status.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 355 | 346 | 349
Score on a scale | 5.2 (0.52) | 5.7 (0.51) | 4.4 (0.51)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.4, 95% CI 2-sided [-1.74 to 0.85]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.8, 95% CI 2-sided [-0.48 to 2.11]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.3, 95% CI 2-sided [-0.04 to 2.56]

21. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Physical Functioning Domain Score at Month 6
Description: SF-36v2 acute is a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 10 items of the physical functioning scale represent levels and kinds of limitations between extremes of physical activities, including lifting and carrying groceries; climbing stairs; bending, kneeling, or stooping; walking moderate distances; self-care limitations. The physical functioning items capture the presence and extent of physical limitations using a 3-level response continuum. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher physical functioning domain score represents better physical functioning.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 348 | 349
Score on a scale | 6.4 (0.52) | 7.3 (0.52) | 7.3 (0.52)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.9, 95% CI 2-sided [-2.22 to 0.39]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.9, 95% CI 2-sided [-2.19 to 0.42]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.0, 95% CI 2-sided [-1.27 to 1.34]

22. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Role Physical Domain Score at Month 6
Description: SF-36v2 acute is a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 4-item role physical scale covers an array of physical health-related role limitations, including: a) limitations in the kind of work or other usual activities; b) reductions in the amount of time spent on work or other usual activities; c) difficulty performing work or other usual activities; and d) accomplishing less. Items in the role physical scale are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher role physical domain score represents better role physical functioning.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 347 | 350
Score on a scale | 6.7 (0.47) | 7.0 (0.47) | 6.3 (0.47)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.3, 95% CI 2-sided [-1.52 to 0.87]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.4, 95% CI 2-sided [-0.80 to 1.58]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.7, 95% CI 2-sided [-0.47 to 1.91]

23. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Bodily Pain Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The bodily pain scale comprises of 2 items pertaining to the intensity of bodily pain and extent of interference with normal work activities. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher bodily pain domain score represents less bodily pain.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 348 | 350
Score on a scale | 8.2 (0.48) | 10.3 (0.48) | 9.9 (0.48)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -2.0, 95% CI 2-sided [-3.25 to -0.80]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -1.7, 95% CI 2-sided [-2.91 to -0.47]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [-0.89 to 1.55]

24. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, General Health Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The general health scale consists of 5 items including a rating of health and 4 items addressing the respondent's view and expectations of his or her health. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher general health domain score represents better general health perceptions.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 347 | 350
Score on a scale | 5.1 (0.44) | 6.3 (0.44) | 5.4 (0.44)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -1.2, 95% CI 2-sided [-2.27 to -0.05]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.3, 95% CI 2-sided [-1.40 to 0.82]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.9, 95% CI 2-sided [-0.25 to 1.98]

25. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Vitality Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 4-item measure of vitality captures a broad range of subjective evaluations of well-being from feelings of tiredness and being worn out to feeling full of energy all or most of the time. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher vitality domain score represents better vitality.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 348 | 350
Score on a scale | 5.6 (0.48) | 6.1 (0.47) | 5.7 (0.47)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.5, 95% CI 2-sided [-1.71 to 0.68]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = -0.1, 95% CI 2-sided [-1.33 to 1.05]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.4, 95% CI 2-sided [-0.83 to 1.57]

26. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Social Functioning Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 2-item social functioning scale assesses health-related effects on quantity and quality of social activities. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher social functioning domain score represents better social functioning.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 348 | 350
Score on a scale | 6.3 (0.52) | 7.2 (0.52) | 6.2 (0.52)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.9, 95% CI 2-sided [-2.20 to 0.45]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.2, 95% CI 2-sided [-1.13 to 1.51]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.1, 95% CI 2-sided [-0.26 to 2.39]

27. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Role Emotional Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 3-item role emotional scale assesses mental health-related role limitations in terms of a) time spent in work or other usual activities; b) amount of work or activities accomplished; c) care with which work or other activities were performed. All 3 items are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher role emotional domain score represents better role emotional functioning.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 347 | 350
Score on a scale | 6.7 (0.58) | 7.7 (0.58) | 6.0 (0.58)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -1.1, 95% CI 2-sided [-2.54 to 0.39]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.7, 95% CI 2-sided [-0.76 to 2.16]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.8, 95% CI 2-sided [0.30 to 3.24]

28. Secondary Outcome: Change From Baseline in the SF-36 Health Survey, Mental Health Domain Score at Month 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 5-item mental health scale includes 1 or more items from each of 4 major mental health dimensions: anxiety, depression, loss of behavioral/emotional control, and psychological well-being. All items are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based scores for both the SF-36 v2 and SF-36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher mental health domain score represents better mental health functioning.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 356 | 348 | 350
Score on a scale | 5.3 (0.52) | 5.5 (0.52) | 5.0 (0.52)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.2, 95% CI 2-sided [-1.55 to 1.08]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.3, 95% CI 2-sided [-1.01 to 1.62]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 0.5, 95% CI 2-sided [-0.78 to 1.86]

29. Secondary Outcome: Change From Baseline in the Work Productivity and Activity Impairment (WPAI) Questionnaire at Month 6
Description: The WPAI: Rheumatoid Arthritis is a 6 item questionnaire that is specific for rheumatoid arthritis and yields four types of scores: absenteeism, presenteesism (impairment at work/reduced job effectiveness), work productivity loss and activity impairment. WPAI outcomes are expressed as impairment percentages ranging from 0 to 100, with higher numbers indicating greater impairment and less productivity.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Percentage of impairment
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 341 | 343
Percentage of impairment
  Work hours missed due to problems | -2.62 (0.717) | -2.19 (0.700) | -1.75 (0.741)
  Work hours missed other reason | 0.14 (1.019) | 0.43 (0.991) | -0.77 (1.059)
  Hours worked in past 7 days | 4.13 (1.729) | -0.82 (1.672) | 1.28 (1.788)
  Problems affecting productivity | -1.94 (0.228) | -2.14 (0.224) | -1.95 (0.232)
  Problem affecting daily activities | -2.24 (0.137) | -2.47 (0.138) | -2.24 (0.139)
  % work time missed due to health | -4.51 (1.790) | -3.41 (1.794) | -1.87 (1.831)
  % impairment while working due to health | -19.38 (2.276) | -21.44 (2.235) | -19.52 (2.320)
  % overall work impairment due to health | -20.16 (2.663) | -22.27 (2.638) | -21.87 (2.710)
  % activity impairment due to health | -22.36 (1.375) | -24.74 (1.383) | -22.45 (1.394)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Work hours missed due to problems; Test type: Superiority or Other; LS mean difference = -0.43, 95% CI 2-sided [-2.279 to 1.427]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Work hours missed due to problems; Test type: Superiority or Other; LS mean difference = -0.87, 95% CI 2-sided [-2.783 to 1.044]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Work hours missed due to problems; Test type: Superiority or Other; LS mean difference = -0.44, 95% CI 2-sided [-2.349 to 1.462]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Work hours missed other reason; Test type: Superiority or Other; LS mean difference = -0.29, 95% CI 2-sided [-2.928 to 2.346]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Work hours missed other reason; Test type: Superiority or Other; LS mean difference = 0.90, 95% CI 2-sided [-1.832 to 3.640]
Statistical Analysis 6: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Work hours missed other reason; Test type: Superiority or Other; LS mean difference = 1.20, 95% CI 2-sided [-1.520 to 3.911]
Statistical Analysis 7: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Hours worked in past 7 days; Test type: Superiority or Other; LS mean difference = 4.95, 95% CI 2-sided [0.520 to 9.370]
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Hours worked in past 7 days; Test type: Superiority or Other; LS mean difference = 2.85, 90% CI 2-sided [-1.736 to 7.430]
Statistical Analysis 9: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Hours worked in past 7 days; Test type: Superiority or Other; LS mean difference = -2.10, 95% CI 2-sided [-6.650 to 2.454]
Statistical Analysis 10: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Problems affecting productivity; Test type: Superiority or Other; LS mean difference = 0.21, 95% CI 2-sided [-0.373 to 0.786]
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Problems affecting productivity; Test type: Superiority or Other; LS mean difference = 0.01, 95% CI 2-sided [-0.578 to 0.607]
Statistical Analysis 12: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Problems affecting productivity; Test type: Superiority or Other; LS mean difference = -0.19, 95% CI 2-sided [-0.784 to 0.400]
Statistical Analysis 13: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Problem affecting daily activities; Test type: Superiority or Other; LS mean difference = 0.24, 95% CI 2-sided [-0.112 to 0.587]
Statistical Analysis 14: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Problem affecting daily activities; Test type: Superiority or Other; LS mean difference = 0.01, 95% CI 2-sided [-0.341 to 0.357]
Statistical Analysis 15: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Problem affecting daily activities; Test type: Superiority or Other; LS mean difference = -0.23, 95% CI 2-sided [-0.582 to 0.122]
Statistical Analysis 16: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; % work time missed due to health; Test type: Superiority or Other; LS mean difference = -1.10, 95% CI 2-sided [-5.748 to 3.553]
Statistical Analysis 17: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; % work time missed due to health; Test type: Superiority or Other; LS mean difference = -2.64, 95% CI 2-sided [-7.339 to 2.067]
Statistical Analysis 18: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; % work time missed due to health; Test type: Superiority or Other; LS mean difference = -1.54, 95% CI 2-sided [-6.283 to 3.207]
Statistical Analysis 19: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; % impairment while working due to health; Test type: Superiority or Other; LS mean difference = 2.07, 95% CI 2-sided [-3.726 to 7.858]
Statistical Analysis 20: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; % impairment while working due to health; Test type: Superiority or Other; LS mean difference = 0.15, 95% CI 2-sided [-5.777 to 6.068]
Statistical Analysis 21: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; % impairment while working due to health; Test type: Superiority or Other; LS mean difference = -1.92, 95% CI 2-sided [-7.839 to 3.998]
Statistical Analysis 22: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; % overall work impairment due to health; Test type: Superiority or Other; LS mean difference = 2.11, 95% CI 2-sided [-4.664 to 8.877]
Statistical Analysis 23: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; % overall work impairment due to health; Test type: Superiority or Other; LS mean difference = 1.71, 95% CI 2-sided [-5.164 to 8.580]
Statistical Analysis 24: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; % overall work impairment due to health; Test type: Superiority or Other; LS mean difference = -0.40, 95% CI 2-sided [-7.307 to 6.510]
Statistical Analysis 25: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; % activity impairment due to health; Test type: Superiority or Other; LS mean difference = 2.38, 95% CI 2-sided [-1.118 to 5.873]
Statistical Analysis 26: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; % activity impairment due to health; Test type: Superiority or Other; LS mean difference = 0.08, 95% CI 2-sided [-3.411 to 3.573]
Statistical Analysis 27: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; % activity impairment due to health; Test type: Superiority or Other; LS mean difference = -2.30, 95% CI 2-sided [-5.818 to 1.225]

30. Secondary Outcome: Change From Baseline in the EuroQol European Quality of Life-5 Dimensions (EuroQol EQ-5D) at Month 6
Description: The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). This profile of scores across the 5-dimensions (e.g. 11231, 33212, etc.) is transformed into a single health utility score using a formula developed by the EuroQol Group that applies country specific preference weights. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. The VAS component rated the current health state on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicating a better health state.
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 348 | 351
Units on a scale
  Utility score | 0.20 (0.013) | 0.22 (0.013) | 0.22 (0.013)
  Mobility score | -0.29 (0.027) | -0.26 (0.027) | -0.28 (0.027)
  Self-care score | -0.27 (0.028) | -0.33 (0.028) | -0.32 (0.028)
  Usual activities score | -0.24 (0.029) | -0.26 (0.029) | -0.30 (0.029)
  Pain/discomfort score | -0.32 (0.026) | -0.34 (0.026) | -0.37 (0.026)
  Anxiety/depression score | -0.21 (0.029) | -0.24 (0.029) | -0.22 (0.029)
  VAS score | 20.84 (1.100) | 20.98 (1.100) | 19.61 (1.100)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Utility score; Test type: Superiority or Other; LS mean difference = -0.02, 95% CI 2-sided [-0.057 to 0.011]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Utility score; Test type: Superiority or Other; LS mean difference = -0.02, 95% CI 2-sided [-0.054 to 0.013]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Utility score; Test type: Superiority or Other; LS mean difference = 0.00, 95% CI 2-sided [-0.031 to 0.036]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Mobility score; Test type: Superiority or Other; LS mean difference = -0.03, 95% CI 2-sided [-0.098 to 0.042]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Mobility score; Test type: Superiority or Other; LS mean difference = -0.01, 95% CI 2-sided [-0.079 to 0.060]
Statistical Analysis 6: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Mobility score; Test type: Superiority or Other; LS mean difference = 0.02, 95% CI 2-sided [-0.051 to 0.089]
Statistical Analysis 7: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Self-care score; Test type: Superiority or Other; LS mean difference = 0.06, 95% CI 2-sided [-0.014 to 0.127]
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Self-care score; Test type: Superiority or Other; LS mean difference = 0.04, 95% CI 2-sided [-0.027 to 0.114]
Statistical Analysis 9: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Self-care score; Test type: Superiority or Other; LS mean difference = -0.01, 95% CI 2-sided [-0.083 to 0.058]
Statistical Analysis 10: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Usual activities score; Test type: Superiority or Other; LS mean difference = 0.01, 95% CI 2-sided [-0.062 to 0.084]
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Usual activities score; Test type: Superiority or Other; LS mean difference = 0.06, 95% CI 2-sided [-0.018 to 0.129]
Statistical Analysis 12: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Usual activities score; Test type: Superiority or Other; LS mean difference = 0.04, 95% CI 2-sided [-0.029 to 0.118]
Statistical Analysis 13: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Pain/discomfort score; Test type: Superiority or Other; LS mean difference = 0.03, 95% CI 2-sided [-0.041 to 0.091]
Statistical Analysis 14: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Pain/discomfort score; Test type: Superiority or Other; LS mean difference = 0.05, 95% CI 2-sided [-0.015 to 0.116]
Statistical Analysis 15: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Pain/discomfort score; Test type: Superiority or Other; LS mean difference = 0.03, 95% CI 2-sided [-0.041 to 0.091]
Statistical Analysis 16: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Anxiety/depression score; Test type: Superiority or Other; LS mean difference = 0.03, 95% CI 2-sided [-0.046 to 0.103]
Statistical Analysis 17: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Anxiety/depression score; Test type: Superiority or Other; LS mean difference = 0.01, 95% CI 2-sided [-0.066 to 0.083]
Statistical Analysis 18: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Anxiety/depression score; Test type: Superiority or Other; LS mean difference = -0.02, 95% CI 2-sided [-0.094 to 0.055]
Statistical Analysis 19: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; VAS score; Test type: Superiority or Other; LS mean difference = -0.14, 95% CI 2-sided [-2.934 to 2.648]
Statistical Analysis 20: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; VAS score; Test type: Superiority or Other; LS mean difference = 1.23, 95% CI 2-sided [-1.556 to 4.016]
Statistical Analysis 21: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; VAS score; Test type: Superiority or Other; LS mean difference = 1.37, 95% CI 2-sided [-1.425 to 4.171]

31. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale Total Score at Month 6
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). The larger the participant's response (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Month 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Number analyzed (Participants) | 357 | 348 | 352
Units on a scale | 7.14 (0.500) | 7.59 (0.498) | 6.07 (0.499)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 5 mg BID + MTX; Test type: Superiority or Other; LS mean difference = -0.45, 95% CI 2-sided [-1.706 to 0.808]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.07, 95% CI 2-sided [-0.178 to 2.325]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + MTX vs Adalimumab 40 mg + MTX; Test type: Superiority or Other; LS mean difference = 1.52, 95% CI 2-sided [0.266 to 2.779]

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent up to at least 28 calendar days after last dose of investigational product. AEs were recorded from the time the subject has taken at least one dose of study treatment through last subject visit.
Description: An event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 5 mg BID + MTX | Adalimumab 40 mg + MTX
Serious Adverse Events (participants affected / at risk) | 35/384 | 27/376 | 24/386
Other Adverse Events (participants affected / at risk) | 51/384 | 72/376 | 69/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=384) | Tofacitinib 5 mg BID + MTX (N=376) | Adalimumab 40 mg + MTX (N=386)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Corneal thinning (Eye disorders) | 1 | 0 | 0
Necrotising retinitis (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 1 | 0
Clostridial sepsis (Infections and infestations) | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Exposure via father (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Enteropathy-associated T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 2
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0
Cellulitis with abscess (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=384) | Tofacitinib 5 mg BID + MTX (N=376) | Adalimumab 40 mg + MTX (N=386)
Nasopharyngitis (Infections and infestations) | 22 | 16 | 18
Upper respiratory tract infection (Infections and infestations) | 25 | 37 | 29
Alanine aminotransferase increased (Investigations) | 8 | 23 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Investigators will, on request, remove any previously undisclosed Confidential Information (other than the Study results themselves) before disclosure.